CLINICAL TRIAL: NCT05164809
Title: Effect of Monopolar Tungsten Needle Electrodes and Teflon Coated Spatula Electrodes on Blood Loss and Intraoperative Transfusions in Musculoskeletal Tumor Surgery Compared to Conventional Surgical Knives and Stainless-Steel Electrodes
Brief Title: Effect of Electrosurgery on Blood Loss and Intraoperative Transfusions in Musculoskeletal Tumor Surgery
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Muenster (Other)
Responsible Party: Principal Investigator, Jan Puetzler, medical doctor, principal investigator, University Hospital Muenster
Other Study IDs: 202101
Record Dates: First submitted 2021-11-19; First posted 2021-12-21 (Actual); Last update posted 2022-01-18 (Actual); Status verified 2022-01

CONDITIONS: Blood Loss, Surgical; Transfusion Rate; Electrosurgery; Tumororthopaedics
MeSH Terms: conditions — Blood Loss, Surgical; Hyperthermia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Tungsten/Teflon +: Dissection with novel electrodes (Tungsten needle electrode + Teflon coated Spatula electrode)
  Interventions: Device: Application of novel electrodes
- Tungsten/Teflon -: Dissection without novel electrodes (Scalpel + Steel Spatula Electrode)

INTERVENTIONS:
Device: Application of novel electrodes — Application of novel electrodes since 2017 for the dissection of extremity tumors in tumororthopedics
  Groups: Tungsten/Teflon +

SUMMARY:
Resection of malign musculoskeletal tumors and reconstruction with large tumor prostheses often results in relevant blood loss requiring hemodynamic stabilization and transfusion.

The use of novel electrosurgical electrodes is assessed retrospectively regarding the potential to reduce blood loss and the need for transfusions.

DETAILED DESCRIPTION:
Background Resection of malign musculoskeletal tumors and reconstruction with large tumor prostheses often result in relevant blood loss requiring hemodynamic stabilization and transfusion. Since machine autotransfusion is contraindicated in tumor surgery, other measures are necessary to reduce intraoperative blood loss.

Objectives Tungsten needle electrodes can be used to simultaneously cut skin and seal bleeding vessels for superficial dissection. Spatula electrodes coated with Teflon (polytetrafluoroethylene PTFE) are used for coagulation and dissection of deeper tissues. The coating reduces eschar build-up and thus smoke creation compared to conventional stainless-steel electrodes. This study assesses the effect of these novel electrodes on blood loss and transfusion rates.

Methods:

The investigators retrospectively investigate all cases of tumor resection and reconstruction with tumor prostheses that were operated five years before the introduction of the new electrodes (2012-2016) and five years after (2018-2021) by one single surgeon with over 25 years of experience. Data are extracted from digital patient records and analyzed by descriptive statistics and t-test for normally distributed data or Mann-Whitney test in case of non-normal distribution.

ELIGIBILITY:
Inclusion Criteria:

* Patients who received hemipelvectomy, hip disarticulation, or major tumor prosthesis implantation at our hospital between 2010 and 2021
* Operated by one single surgeon

Exclusion Criteria:

- Implantation of a Megaprosthesis without history of tumor

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A defined number of cases is available. All patients with tumor resection and replacement with tumor prosthesis in the orthopedic department at UKM (2012-2016 with conventional dissection instruments and 2018-2021 with novel electrodes) from one single surgeon with over 25 years experience
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-02 (Estimated)

PRIMARY OUTCOMES:
Blood loss | during surgery
  monitored during surgery in the anaesthesiology protocol
Transfusion of red packed blood cells | during surgery
  number of intraoperative units of packed red blood cells
Transfusion of red packed blood cells | 14 days post surgery
  number of intraoperative units of packed red blood cells

SECONDARY OUTCOMES:
post surgical wound drainage | 5 days post surgey
  assessed via recorded volume

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No
No IPD will be shared

REFERENCES:
- [Derived] Puetzler J, Steinbicker AU, Santel J, Deventer N, Jahn M, Zarbock A, Gosheger G, Schulze M, Jenke DJ. Blood-saving dissection with monopolar tungsten needle electrodes and Teflon-coated spatula electrodes in tumor orthopedics. J Orthop Traumatol. 2023 May 15;24(1):22. doi: 10.1186/s10195-023-00704-8. PMID 37188890